CLINICAL TRIAL: NCT06859931
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Clinical Trial Evaluating the Efficacy and Safety of TQB3702 Tablets in Patients With Systemic Lupus Erythematosus
Brief Title: Clinical Trial of TQB3702 Tablets in Subjects With Systemic Lupus Erythematosus (SLE)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB3702-II-01
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-12

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TQB3702 Tablets (Experimental): Administer orally on an empty stomach, once daily, for 24 consecutive weeks.
  Interventions: Drug: TQB3702 Tablets
- TQB3702 Tablets+TQB3702 Placebo (Experimental): Administer orally on an empty stomach, once daily, for 24 consecutive weeks. Placebo was administered orally once a day for 24 weeks.
  Interventions: Drug: TQB3702 Tablets+TQB3702 Placebo
- TQB3702 Placebo (Placebo Comparator): Placebo was administered orally once a day for 24 weeks.
  Interventions: Drug: TQB3702 Placebo

INTERVENTIONS:
Drug: TQB3702 Tablets — TQB3702 is a selective kinase inhibitor.
  Arms: TQB3702 Tablets
Drug: TQB3702 Tablets+TQB3702 Placebo — TQB3702 is a selective kinase inhibitor； A placebo is a simulated drug whose physical properties, such as appearance, size, color, dosage form, weight, taste, and odor are substantially the same as the test drug, but cannot contain the active ingredients of the test drug.
  Arms: TQB3702 Tablets+TQB3702 Placebo
Drug: TQB3702 Placebo — TQB3702 Placebo without drug substance.
  Arms: TQB3702 Placebo

SUMMARY:
TQB3702 is a selective kinase inhibitor. This is a Phase II clinical study aimed at evaluating the efficacy and safety of TQB3702 tablets in patients with systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participate in the study and sign the informed consent;
* Male and female, ≥18 years old and ≤70 years old (subject to the date of signing the informed consent);
* The diagnosis meets the classification criteria of SLE established by the International Clinical Collaboration on Lupus Research (SLICC) in 2012 and has been in place for at least 6 months (Appendix 16), excluding drug-related lupus;
* Meet the Systemic lupus erythematosus disease activity index-2K score requirements
* Positive for one or more of the following antibodies: positive for anti-nuclear antibodies (ANA titers greater than or equal to 1:80 by immunofluorescence) and/or positive for anti-DSDNA antibodies and/or positive for anti-Smith(anti-SM);
* Subjects were receiving standard treatment for SLE and had received treatment for at least 3 months prior to randomization. Standard therapeutic doses of SLE were stable for at least 30 days and glucocorticoids were stable for at least 2 weeks prior to initial administration. The standard treatment for SLE may be corticosteroids, and/or antimalarial drugs, and/or immunosuppressants
* At the time of screening, if the subject is taking an angiotensin-converting enzyme inhibitor or an angiotensin-II receptor blocker or a non-steroidal anti-inflammatory drug (NSAID) orally, it must be at least 2 weeks since the pre-screening dose stabilized;
* Subjects must stop all opioids at least 1 week before the first dose;
* Fertile subjects must consent to and commit to using a medically accepted form of contraception throughout the study period and for at least 6 months after the final trial drug administration.

Exclusion Criteria:

* Subjects who are pregnant or lactating, or who plan to have a child in the 12 months prior to the first dosing.
* Severe lupus nephritis within 30 days prior to initial administration;
* Central nervous system diseases caused by SLE or not caused by SLE in the 12 months before the first dose;
* Current or past autoimmune diseases other than SLE
* There is an active and uncontrolled infection, or an infection that has recently required intravenous anti-infective therapy, or is currently being treated for any chronic infection
* Subjects whose chest radiology within 6 months prior to screening indicates active tuberculosis
* Have active hepatitis, or hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive + hepatitis B virus (HBV) DNA positive, or hepatitis C virus (HCV) RNA positive; Or a history of human immunodeficiency virus (HIV) infection, or a positive HIV serological result at screening; The specific antibody of Treponema pallidum was positive and the confirmatory test was positive. If HBV core antibody is positive but HBV-DNA is negative, HBV-DNA should be monitored once every 3 months.
* Herpes or shingles infection, or a history of disseminated/complicated shingles in the 12 weeks prior to screening;
* Cardiovascular and cerebrovascular abnormalities;
* Have a lung disease that the investigator determines is not suitable for participation in the study
* Subjects with a history or suspected demyelinating disease of the central nervous system;
* Subjects with a history of or suspected demyelinating disease of the central nervous system;
* Subjects with any type of active malignancy or with a history of malignancy;
* Have a history of vital organ transplantation or hematopoietic stem cell/bone marrow transplantation;
* The subject has any medical condition that may affect the absorption of oral medications (e.g., bariatric/obesity surgery, or the subject is unable to take oral medications;
* Previous use of specific drugs;
* Patients who underwent plasma replacement within 12 weeks prior to initial administration or treated with human immunoglobulin 4 weeks prior to initial administration;
* Cyclophosphamide had been used within 3 months before the first dose;
* Rituximab or any other B-cell depletion therapy within 6 months prior to initial administration;
* Use Beliuzumab, Taitacept, tumor necrosis factor (TNF) antagonists, or other biologics before initial administration unless the elution time is met, as specified in Appendix 17;
* Participants who have suffered a major trauma, fracture, or surgical procedure in the 4 weeks prior to screening, or who are expected to require major surgical procedures during the study period;
* Participants who received live attenuated vaccine within 28 days before the start of study treatment, inactivated vaccine within 7 days, or planned vaccination during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
SLE response index -4 (SRI-4) | Baseline to week 24
  ≥4 point reduction from baseline in systemic lupus erythematosus disease activity index 2000 (SLEDAI-2k) score and no new the British Isles Lupus Assessment Group (BILAG) A score and no more than one new BILAG B organ domain score compared with baseline and no worsening in Physician Global Assessment (PGA) (<0.3 points increase from baseline).

SECONDARY OUTCOMES:
SLE response index -4 (SRI-4) | Baseline to weeks 4 and 12
  ≥4 point reduction from baseline in SLEDAI-2k score AND no new BILAG A score and no more than one new BILAG B organ domain score compared with baseline AND no worsening in PGA (<0.3 points increase from baseline)
SLE response index -6 (SRI-6) | Baseline to weeks 4, 12, and 24
  ≥6 point reduction from baseline in SLEDAI-2k score AND no new BILAG A score and no more than one new BILAG B organ domain score compared with baseline AND no worsening in PGA (<0.3 points increase from baseline)
SLE Disease Activity Index -2000 score | Baseline to weeks 4, 12, and 24
  A tool for assessing disease activity in systemic lupus erythematosus (SLE), with a score based primarily on whether a patient develops clinical symptoms within 28 days.
  The higher the score, the higher the patient's disease activity.
Cutaneous lupus erythematosus Area and Severity Index (CLASI score) | Baseline to weeks 4, 12, and 24
  A useful tool for assessing skin activity in patients with lupus erythematosus. The higher the score, the higher the patient's disease activity.
Number of active (tender + swollen) joints | Baseline to weeks 4, 12, and 24
  Changes in the number of joints subject moves (tenderness + swelling)
Medical Outcomes Study 36-Item Summary Health Survey (SF-36) | Baseline to weeks 12
  Changes in 36 summary health surveys in the Medical Outcomes Study. The higher the score, the better the patient's self-reported quality of life.
The change of Anti double-stranded DeoxyriboNucleic Acid(ds-DNA) antibody Anti-dsdna antibody and antinuclear antibody (ANA) | Baseline to weeks 4, 12, and 24
  The change of anti-dsDNA antibody value and ANA value
Changes in Complement 3 (C3) values and Complement 4 (C4) values | Baseline to weeks 4, 12, and 24
  Changes in C3 values and C4 values
Immunoglobulin G (IgG), Immunoglobulin M (IgM), Immunoglobulin A (IgA) levels | Baseline to weeks 4, 12, and 24
  Changes of IgG, IgM and IgA levels.
Cytokine expression levels | Baseline to weeks 4, 12, and 24
  Changes in cytokine expression levels
Total B cell count | Baseline to weeks 4, 12, and 24
  Changes in total B cell count
Erythrocyte sedimentation rate (ESR) | Baseline to weeks 4, 12, and 24
  Changes in erythrocyte sedimentation rate
Frequency of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The occurrence of all adverse medical events after the first injection.
Severity of adverse event (AE) | From the date of signing the informed consent to 28 days after the last dosing or a new anti-tumor treatment, whichever comes first.
  The severity of all adverse medical events after the first injection.
Peak time (Tmax) | 1, 84, 112, 140 and 168 Days
  Peak time (Tmax)
Target occupancy | Day 1, 14 and 168
  The extent to which the drug occupies the target on the cell surface
Peak concentration (Cmax) | 1, 84, 112, 140 and 168 Days
  Peak concentration (Cmax)
Area under the blood drug concentration time curve (AUC0-24h, AUC0-t, AUC0- ∞), | 1, 84, 112, 140 and 168 Days
  Area under the blood drug concentration time curve (AUC0-24h, AUC0-t, AUC0- ∞),
Apparent volume of distribution (Vd/F) | 1, 84, 112, 140 and 168 Days
  Apparent volume of distribution (Vd/F)
Plasma clearance rate (CL/F) | 1, 84, 112, 140 and 168 Days
Plasma elimination half-life (t1/2) | 1, 84, 112, 140 and 168 Days
  Plasma elimination half-life (t1/2)
Steady-state peak time (Tmax, ss) | 1, 84, 112, 140 and 168 Days
  Steady-state peak time (Tmax, ss)
Steady-state peak concentration (Cmax, ss) | 1, 84, 112, 140 and 168 Days
  Steady-state peak concentration (Cmax, ss)
Steady-state trough concentration (Cmin, ss) | 1, 84, 112, 140 and 168 Days
  Steady-state trough concentration (Cmin, ss)
Average steady-state blood drug concentration (Cav, ss) | 1, 84, 112, 140 and 168 Days
  Average steady-state blood drug concentration (Cav, ss)
Area under the steady-state blood drug concentration time curve (AUCss) | 1, 84, 112, 140 and 168 Days
  Area under the steady-state blood drug concentration time curve (AUCss)
Accumulation ratio (Rac) | 1, 84, 112, 140 and 168 Days
  Accumulation ratio (Rac)
Volatility (DF) | 1, 84, 112, 140 and 168 Days
  Volatility (DF)

CONTACTS AND LOCATIONS:
Locations (37):
- China (37):
  - The First Affilliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The People's Hospital of Gansu Province, Lanzhou, Gansu
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen second people's hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hebei petro China central hospital, Langfang, Hebei
  - The second hospital of hebei medical university, Shijiazhuang, Heibei
  - Puyang Oilfield General Hospital, Puyang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shiyan People's Hospital, Shiyan, Hubei
  - Huazhong University of Science and Technology Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Third Hospital of Central South University, Changsha, Hunan
  - Shaoyang Central Hospital, Shaoyang, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Shenjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Hospital Affiliated to the Army Medical University, Xi'an, Shaanxi
  - Affiliated hospital of Shandong Academy of Medical Sciences, Jinan, Shandong
  - Shanghai Jiao Tong University School of Medicine，Renji Hospital, Shanghai, Shanghai Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - First Hospital of Shangxi Medical University, Taiyuan, Shanxi
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Mianyang central hispital, Mianyang, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Third People's Hospital of Yunnan Province, Kunming, Yunnan
  - Pu'er People's Hospital, Pu'er, Yunnan
  - Taizhou Central Hospital（Taizhou University Hospital）, Taizhou, Zhejiang
  - The 1th School of Medicine,School of Information and Engineering,The 1th Affiliated Hospital of WMU, Wenzhou, Zhejiang
  - Wenzhou People's Hospital, Wenzhou, Zhejiang